CLINICAL TRIAL: NCT02509364
Title: Study of the Etiology and Immunological Pathogenesis in Acute Exacerbation of Idiopathic Pulmonary Fibrosis (AE-IPF)
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Shanghai Pulmonary Hospital, Shanghai, China (Other)
Responsible Party: Principal Investigator, Huiping Li, Chief Physician, Shanghai Pulmonary Hospital, Shanghai, China
Other Study IDs: SPH150715
Record Dates: First submitted 2015-07-20; First posted 2015-07-28 (Estimated); Last update posted 2015-07-28 (Estimated); Status verified 2015-07

CONDITIONS: Interstitial Lung Diseases
Keywords: AE-IPF
MeSH Terms: conditions — Lung Diseases, Interstitial

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Sputum, throat swab, BALF and blood will be collected in this study.

GROUPS / COHORTS (3):
- AE-IPF: Diagnosis criteria for AE-IPF:
  * Diagnosed IPF patient experiences unexplained dyspnea within 1 month
  * With objective evidence of hypoxia and new onset of pulmonary infiltration based on imaging examination
  * With other diagnosis like pulmonary embolism, pneumothorax or heart failure excluded.
  Interventions: Other: No intervention
- Stable-IPF: Diagnosis criteria for Stable-IPF:
  * Exclusion of other known causes of ILDs
  * Presence of a usual interstitial pneumonitis (UIP) pattern on high-resolution computed tomography (HRCT)
  * Specific combinations of HRCT and surgical lung biopsy pattern in patients subjected to surgical lung biopsy.
  Interventions: Other: No intervention
- Health control: Healthy volunteer
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention

SUMMARY:
Idiopathic pulmonary fibrosis (IPF) is a highly heterogeneous and lethal pathological process with limited therapeutic options, which is the most common and severe of the idiopathic interstitial pneumonias (IIPs). During the past 20 years, the incidence of IPF increased significantly. Most of IPF patients show a median survival time of 2-3 years after diagnosis. Five-year survival rate is 30%-50%. It's difficult to diagnose in the early stage of IPF. Once the patients go to hospital, it's already in the late stage. Now there is no effective therapy except lung transplant for IPF in clinical application.

Acute exacerbation of idiopathic pulmonary fibrosis (AE-IPF) is a fatal condition with high mortality (over 80%). Its etiology and pathogenesis remain unknown. There is a lack of effective treatment for it. Based on the investigators' long-term clinical observation, most cases of AE-IPF initially got "common cold" and had coryza, more cough, nasal obstruction，rhinorrhea, sore throat, some patients had fever, headache, and etc. Some of these patients' condition developed very rapidly and then became very severe similar to the situation of acute respiratory distress syndrome (ARDS). Why these AE-IPF patients were so hypersensitive to "cold"? What were the immunologic and pathological mechanisms of their lung lesions after patients exposed to "common cold"? How to effectively offer interventional treatment for AE-IPF? All the above questions are yet to be explained clearly.

In the investigators' previous retrospective study, the investigators found that there were some obviously imbalanced immune responses in IPF patients, including increased cluster of differentiation 4 (CD4) T cell population, immunoglobulin and complements. The investigators also found highly expressed inflammatory cytokines (IL-17, MIG and IL-9) and high detection rates of pathogens in AE-IPF patients, especially serum immunoglobulin M (IgM) antibody of some respiratory virus. These findings provide a strong suggestion that there are some imbalance of immunologic function in IPF and there are relationship between AE-IPF and infection, especially "Cold" virus infection might be a key trigger for AE-IPF.

DETAILED DESCRIPTION:
IPF has become the focus of study in the area of pulmonary fibrosis, accounting for over 25% of all interstitial lung diseases (ILD) 1 and over 60% of all idiopathic interstitial pneumonia (IIP). The past 20 years have observed the remarkable tendency of increase of IPF incidence, accompanied by only 2-3 years of medium survival after diagnosis and 30-50% of 5-year survival2. Due to limited diagnosis method at early stage of the disease, the patients are most likely diagnosed only when they reach middle or late stage. Other issue is lack of effective treatment, except for lung transplantation. Most of the deaths are caused by acute exacerbation, which is defined by clinicians as acute exacerbation of IPF (AE-IPF) and characterized by the rapid deterioration during relatively stable period of IPF (Stable-IPF). Exacerbation may occur at all stages of IPF development (see the below figure) and is accompanied by hazardous and quick development, high mortality and very poor prognosis.

The incidence and mortality of AE-IPF varies in different studies. Kubo etc. reported that acute exacerbation occurs within 3 years in around 57% of IPF patients, with the mortality of 53%. Study by Kim etc. show that the mortality of AE-IPF reaches 78%. Study by Song etc.demonstrated that the incidence of acute exacerbation of IPF is 35.4%, with over 50% of in-hospital morality, 56% of 1-year mortality and 18.4% of 3-year mortality. Other studies showed that 1-year post-exacerbation mortality is nearly 100%. Data based on the 178 in-hospital IPF patients in the investigators' department during the latest 4 years showed that 58% (102/178) of those patients experienced acute exacerbation at certain stage of disease, with 70 deaths occurred. Among those deaths, 56 cases (83%) were caused by acute exacerbation. It is clear that the high incidence and mortality of AE-IPF is the most essential factors impacting the survival and quality of life of IPF patients, therefore lead to the poor prognosis of IPF.

Hypothesis and key scientific questions Based on analysis above, the investigators propose the following hypothesis: certain level of immunological imbalance exists in those relatively stable IPF patients, making them susceptible to infection by various pathogens. Once infected, especially by viruses (e.g. common cold related viruses), AE-IPF can be quickly triggered, leading to ARDS-like reaction. To validate this hypothesis, four key scientific questions need to be answered by studies with scrupulous design: 1) what are the characteristic changes of immunological function in IPF/AE-IPF patients so as to make the patients more susceptible to common cold viruses? 2) What kind of pathogens, especially those common cold viruses, are the key triggering factors during the development of AE-IPF? 3) What kind of inflammatory cascade reaction occurs in AE-IPF leading to ARDS-like prompt development of pulmonary inflammation? Key research direction and scientific rationale In order to address the key scientific questions above, the investigators will conduct comprehensive studies based on detailed screen and analysis of large amount of clinical cases, integrated research methods in such areas as immunology, molecular, cytology and animal model, as well as high throughput data collection and big data analysis: 1) Extensive screening and identification of those pathogens closely related with AE-IPF; 2) Comprehensive analysis of the change of immunology function, focusing on the pathological-physiological alteration in virus induced immunologic imbalance in IPF, as well as the characteristic changes in relevant cytological signal transduction, so as to identify important AE-IPF bio-markers and explain the pathological molecular mechanism and network of ARDS-like inflammatory cascade reaction, which will be significant efforts in terms of prevention of AE-IPF, reduction of mortality, improvement of quality of life, delaying of disease progression and increase of survival.

Similar clinical deterioration like AE-IPF will also occur in almost all the other types of pulmonary fibrosis, especially connective tissue disease-ILD (CTD-ILD), nonspecific interstitial pneumonia (NSIP), drug induced ILD, fibrotic allergic pneumonia and cryptogenic organizing pneumonia (COP) etc. Therefore, this program will also provide insight into the basic research and clinical management of acute exacerbation of other interstitial lung diseases, which is one common problem extensively exists in the area of interstitial lung disease and the key factor in terms of improving patients' quality of life and survival.

ELIGIBILITY:
Inclusion Criteria:

Clinical diagnosis of IPF:

* Exclusion of other known causes of ILDs
* Presence of a UIP pattern on HRCT
* Specific combinations of HRCT and surgical lung biopsy pattern in patients subjected to surgical lung biopsy.

Clinical diagnosis of AE-IPF:

* Diagnosed IPF patient experiences unexplained dyspnea within 1 month
* With objective evidence of hypoxia and new onset of pulmonary infiltration based on imaging examination
* With other diagnosis like pulmonary embolism, pneumothorax or heart failure excluded.

Exclusion Criteria:

-Not applicable.

Ages: 54 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subject cohorts: Cohort 1: Stable IPF group (n>150); Cohort 2: AE-IPF group (n>50); Cohort 3: healthy control group (n>100). All the IPF patients have been enrolled according to relevant diagnosis criteria. The criteria of AE-IPF include: diagnosed IPF patient experiences unexplained dyspnea within 1 month, with objective evidence of hypoxia and new onset of pulmonary infiltration based on imaging examination, and with other diagnosis like pulmonary embolism, pneumothorax or heart failure excluded.Serial observation of the change of pathogens based on at least two times of sample collection. Healthy control group recruits healthy population based on physical exam, with no definite respiratory disease and normal chest X ray results.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2015-08; Primary Completion 2016-12 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
Virus RNA by pathogen test chip and second generation sequencing in AE-IPF | up to 30 weeks
  Testing of pathogen nucleic acid chips:Based on PathGEN® Pathogen Chip Kit (PathGEN Dx, Singapore). Next Generation Sequencing (NGS) has become the powerful tool in pathogen identification based on its rapidness and sensitivity. The final report will provide the species classification of the bacteria and viruses, as well as corresponding designator.
Macrophage phenotype and function | up to 30 weeks
  Subtype and functional testing on phenotype and function of Macrophage cell in IPF/AE-IPF patients.
Dendritic cell (DC) phenotype and function | up to 30 weeks
  Subtype and functional testing on phenotype and function of DC in IPF/AE-IPF patients.
T cell phenotype and function | up to 30 weeks
  Subtype and functional testing on phenotype and function of T cell in IPF/AE-IPF patients.
B cell phenotype and function | up to 30 weeks
  Subtype and functional testing on phenotype and function of B cell in IPF/AE-IPF patients.
Expression of IL-17 in AE-IPF | up to 30 weeks
  The investigators will evaluate the expression of IL-17 by proteomics in IPF/AE-IPF patients.
Expression of MIG in AE-IPF | up to 30 weeks
  The investigators will evaluate the expression of MIG by proteomics in IPF/AE-IPF patients.

CONTACTS AND LOCATIONS:
Overall Officials: Huiping Li, MD,PhD, Principal Investigator — Shanghai Pulmonary Hospital, Tongji University, Shanghai, China
Locations (1):
- Shanghai Pulmonary Hospital, Tongji University, Shanghai, Shanghai Municipality, China